CLINICAL TRIAL: NCT07177430
Title: The Effect of Inspiratory Muscle Training on Respiratory Function, Exercise Tolerance and Core Stability in Children and Adolescents With Idiopathic Scoliosis Undergoing Schroth Therapy.
Brief Title: Inspiratory Muscle Training in Children and Adolescents With Idiopathic Scoliosis Undergoing Schroth Therapy.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wroclaw University of Health and Sport Sciences (Other)
Responsible Party: Principal Investigator, Aleksandra Grudzińska, MSc, Wroclaw University of Health and Sport Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: WroclawUHSS Ethics (22/2025)
Record Dates: First submitted 2025-08-29; First posted 2025-09-17 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Scoliosis Idiopathic
Keywords: Inspiratory Muscle Training; Schroth method; Exercise tolerance; Core stability; Respiratory function
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sham Group (Sham Comparator): IMT (Sham) and Schroth therapy
  Interventions: Device: Inspiratory Muscle Training (Sham)
- IMT Group (Experimental): IMT and Schroth therapy
  Interventions: Device: Inspiratory Muscle Training

INTERVENTIONS:
Device: Inspiratory Muscle Training — Participants will perform inspiratory muscle training using a respiratory muscle trainer. The initial training load will be set at 30% of PImax.
  The intervention will last for 8 weeks and will be carried out 5 days per week, twice daily, in 3 sets of 10 repetitions.
  The training load will be increased in the 2nd, 4th, and 6th week of the program, each time by an additional 10% relative to the initial PImax.
  Arms: IMT Group
Device: Inspiratory Muscle Training (Sham) — The training intervention in the Sham Group will differ from the experimental group only in terms of training load.
  This load will remain constant at 15% PImax, which does not cause any changes in the functioning of the inspiratory muscles.
  All other training parameters will be identical to those in the IMT group.
  Arms: Sham Group

SUMMARY:
This study evaluates the effectiveness of inspiratory muscle training in children and adolescents with idiopathic scoliosis undergoing therapy with the Schroth method.

The intervention- inspiratory muscle training- aims to improve respiratory function, increase exercise tolerance, and strengthen core stability in the participants.

The proposed training may enhance the effectiveness of therapy conducted using the Schroth method and improve participants' performance in activities of daily living.

The project aims to assess the impact of inspiratory muscle training in children and adolescents with idiopathic scoliosis on respiratory system function, exercise tolerance, and core stability.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed idiopathic scoliosis,
* age: 11-16 years (girls after their first period, boys after voice mutation),
* spinal curvature angle > 20° according to Cobb,
* guardian's consent to participate in the study;

Exclusion Criteria:

* chronic respiratory diseases,
* inhalant allergies,
* limited contact with the patient, preventing the examination from being performed;

Ages: 11 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 56 (Estimated)
Dates: Start 2025-10-13 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Pulmonary function test | Baseline and after 8 weeks (post-intervention)
  Assessment of pulmonary ventilation will be performed using pulmonary function testing with a MasterScreen Pneumo spirometer (Jaeger). This examination is non-invasive and performed in accordance with ATS and ERS criteria.
  The data collected for analysis will include the following parameters: vital capacity (VC), forced vital capacity (FVC), forced expiratory volume in one second (FEV1), peak expiratory flow (PEF), maximal expiratory flow at 50% of forced vital capacity (MEF50).
  Unite of measurements: all measurements are taken as a percentage from predicted.
Pulmonary function test (Maximal inspiratory flow at 50% of FVC (MIF50)) | Baseline and after 8 weeks (post-intervention)
  Pulmonary function test will be performed using a MasterScreen Pneumo spirometer (Jaeger). This examination is non-invasive and performed in accordance with ATS and ERS criteria.
  Maximal inspiratory flow at 50% of FVC (MIF50) is expressed in litres per second (l/s).
Pulmonary function test (MEF50/MIF50 ratio) | Baseline and after 8 weeks (post-intervention)
  Pulmonary function test will be performed using a MasterScreen Pneumo spirometer (Jaeger). This examination is non-invasive and performed in accordance with ATS and ERS criteria.
  The MEF50/MIF50 ratio is a dimensionless value (because in this case the MEF50 value is expressed in l/s, similarly to MIF50). This indicator assesses airway patency. It is mainly used for the diagnosis and differentiation of upper airway stenosis.
Measurement of maximal inspiratory and expiratory pressure | Baseline and after 8 weeks (post-intervention)
  Respiratory muscle strength will be assessed by measuring maximal inspiratory and expiratory pressure. The test is non-invasive and will be performed using a pneumatic adapter connected to the tachometer of the device used for pulmonary function testing. The assessment will be conducted in accordance with ATS/ERS guidelines; following the recommended procedure, 5 to 10 measurements will be taken, from which the three highest values will be selected.
  Based on the results of this test, the training parameters for the planned intervention will be determined.
Forced oscillation technique (FOT) | Baseline and after 8 weeks (post-intervention)
  To provide information on the mechanical and elastic properties of the respiratory system, the forced oscillation technique (FOT) will be performed. For this purpose, the Resmon Pro V3 device (MGC Diagnostics®) will be used, employing the built-in pediatric mode that applies an 8 Hz signal frequency. The main parameters analyzed will be resistance (Rrs) and reactance (Xrs).
Six-minute walk test (6MWT) | Baseline and after 8 weeks (post-intervention)
  This test will be used to assess cardiorespiratory fitness. The examination will be conducted in accordance with the American Thoracic Society guidelines for this test. The parameter analyzed will be the distance covered by the participants.
Isokinetic dynamometry (Peak torque) | Baseline and after 8 weeks (post-intervention)
  Isokinetic dynamometry using the Biodex Multi-Joint System will be employed to assess the participants' ability to maintain postural stability in different planes under static and isokinetic conditions.
  Assessed muscle groups responsible for trunk stabilization: trunk flexors (abdominal muscles) and trunk extensors (back muscles).
  The evaluated parameter, peak torque, represents the maximum recorded torque produced by the analyzed muscle group at a specified angular velocity, expressed in newton-meters (N·m).
  Measurements will consist of performing trunk flexion and extension as quickly as possible with maximal force at two angular velocities. A warm-up will be conducted prior to testing. Five maximal trials will be performed, with rest periods between trials. During the trials, participants will be verbally encouraged to exert maximal effort.
Isokinetic dynamometry (Total work) | Baseline and after 8 weeks (post-intervention)
  Isokinetic dynamometry using the Biodex Multi-Joint System will be employed to assess the participants' ability to maintain postural stability in different planes under static and isokinetic conditions.
  Assessed muscle groups responsible for trunk stabilization: trunk flexors (abdominal muscles) and trunk extensors (back muscles).
  Total work is the work performed by the muscles throughout all movements executed during the task. It also allows for the assessment of muscle endurance. This parameter is expressed in joules (J).
  Measurements will consist of performing trunk flexion and extension as quickly as possible with maximal force at two angular velocities. A warm-up will be conducted prior to testing. Five maximal trials will be performed, with rest periods between trials. During the trials, participants will be verbally encouraged to exert maximal effort.
Isokinetic dynamometry (Average power) | Baseline and after 8 weeks (post-intervention)
  Isokinetic dynamometry using the Biodex Multi-Joint System will be employed to assess the participants' ability to maintain postural stability in different planes under static and isokinetic conditions.
  Assessed muscle groups responsible for trunk stabilization: trunk flexors (abdominal muscles) and trunk extensors (back muscles).
  Average power is a parameter calculated by dividing the work performed during a single repetition by the duration of the movement. Its values are expressed in watts (W).
  Measurements will consist of performing trunk flexion and extension as quickly as possible with maximal force at two angular velocities. A warm-up will be conducted prior to testing. Five maximal trials will be performed, with rest periods between trials. During the trials, participants will be verbally encouraged to exert maximal effort.

SECONDARY OUTCOMES:
Physical activity | Before intervention
  Physical activity levels will be assessed using the PAQ-C (Physical Activity Questionnaire for Children) or PAQ-A (Physical Activity Questionnaire for Adolescents). This questionnaire gathers information on the frequency and intensity of physical activities, including sports, outdoor play, and other forms of exercise. Higher scores indicate greater levels of physical activity.

CONTACTS AND LOCATIONS:
Overall Officials: Krystyna Rożek-Piechura, Professor, Study Director — Wroclaw University of Health and Sport Sciences, Poland; Aleksandra Grudzińska, MSc, Principal Investigator — Wroclaw University of Health and Sport Sciences, Poland; Elżbieta Piątek-Krzywicka, PhD, Principal Investigator — Wroclaw University of Health and Sport Sciences, Poland; Anna Badowska, MD, Principal Investigator; Jerzy R Piechura, PhD, Principal Investigator — Wroclaw University of Health and Sport Sciences, Poland; Paulina Okrzymowska, PhD, Principal Investigator — Wroclaw University of Health and Sport Sciences, Poland
Locations (2):
- Poland (2):
  - Centrum Skolioz- Centrum Diagnostyczno-Rehabilitacyjne Promyk Słońca, Wroclaw, Lower Silesian Voivodeship
  - Wroclaw University of Health and Sport Sciences, Wroclaw, Lower Silesian Voivodeship